CLINICAL TRIAL: NCT03860168
Title: PICU Up!:A Pilot Stepped-wedge Trial of a Multicomponent Early Mobility Intervention for Critically Ill Children
Brief Title: PICU Up!: A Pilot Stepped-wedge Trial of a Multicomponent Early Mobility Intervention for Critically Ill Children
Acronym: PICU Up!
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Donaghue Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00199373; 789 (Other: Other)
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness
Keywords: sleep; sedation; early mobilization; acute rehabilitation; delirium
MeSH Terms: conditions — Critical Illness; Delirium

STUDY DESIGN:
Intervention Model Description: The study will be conducted using a pragmatic stepped-wedge cluster randomized trial (RCT) design, with each PICU acting as one cluster. In a traditional stepped-wedge (TSW) design, all clusters begin in the control group and then transition to the intervention group at sequential and randomly assigned periods, facilitating the delivery of a desired intervention to all clusters, in this case, all participating PICUs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PICU Up! pre- and post-implementation (Other): Each unit will begin in the baseline, usual care phase and then be randomized to implement the PICU Up! program during a set time period, followed by the post-implementation phase.
  Interventions: Other: PICU Up!

INTERVENTIONS:
Other: PICU Up! — The PICU Up! intervention is a multifaceted mobility program incorporating the ABCDEF bundle components into routine PICU care through multidisciplinary staff education and a structured pathway to determine a patient's daily mobility goal. PICU Up! was developed by a collaborative multidisciplinary team approach, and the central components include the consultation and involvement of physical therapy/occupational therapy (PT/OT) by PICU Day 3, sleep hygiene promotion and routine delirium screening for all PICU patients utilizing a validated tool.

SUMMARY:
Recent decreases in Pediatric Intensive Care Unit (PICU) mortality rates have been offset by increased morbidity and length of stay for vulnerable young patients. Heavy sedation, bedrest, and delirium contribute to a PICU culture of immobility. While studies in adult ICU patients demonstrate the clinical benefits of early mobilization, fewer than 25% of critically ill children mobilize early in the children's PICU stay. The investigators have demonstrated the safety and feasibility of the 'PICU Up!' Mobility Program, which integrates sleep promotion, delirium prevention, sedation optimization as a bundle to increase mobilization. However, the generalizability and broader impact on patient- and family-centered outcomes is unknown. Therefore, there is an urgent need for trials that blend both clinical effectiveness and implementation research to create a PICU culture of mobility and improve the value of PICU care. The overall objective of the proposed research is to determine the impact of a transdisciplinary and multifaceted early mobility program on clinical outcomes and ICU-acquired morbidities in critically ill children. Additionally, the investigators will identify barriers and facilitators to high-performance bundle adoption.

ELIGIBILITY:
Inclusion Criteria for Participating Units:

* Participating PICUs must be a separate physical space dedicated to the care of critically ill infants and children, with the ability to provide mechanical ventilation.
* Not implemented a PICU mobility protocol and would commit to not implementing a mobility protocol until the randomized time of unit implementation.

Inclusion Criteria for Patients:

All patients admitted to the PICUs regardless of length of stay will receive the unit-based PICU Up! intervention, which includes criteria for no mobilization based on specific clinical factors (i.e. open chest, surgeon request).10 For inclusion in data analysis, patients will be eligible if

* Admitted to the participating PICU ≥ 3 days.

Exclusion Criteria for Patients:

* Patients with an active do-not-resuscitate (DNR) order will be excluded.

Ages: 0 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2500 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation (days) | 28 days
  Defined as the number of days of mechanical ventilation through an endotracheal tube during the first 28 days of PICU admission.

SECONDARY OUTCOMES:
PICU length of stay (days) | 28 days
Hospital length of stay (days) | 28 days
Proportion of patients receiving out-of-bed mobility before PICU Day 28 | 28 days
Number of patients discharged directly to home from the PICU | 28 days
Number of patients discharged from the hospital to a place other than home | 28 days
  Number of patients discharged from the hospital to a place other than home (rehabilitation facility) if previous residence was home
Incidence of venous thromboembolism | 28 days
Incidence of pressure injury | 28 days
Cumulative exposure to opioids (mg/kg) through PICU Day 28 | 28 days
Cumulative exposure to benzodiazepines (mg/kg) through PICU Day 28 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Sapna R Kudchadkar, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Wieczorek B, Ascenzi J, Kim Y, Lenker H, Potter C, Shata NJ, Mitchell L, Haut C, Berkowitz I, Pidcock F, Hoch J, Malamed C, Kravitz T, Kudchadkar SR. PICU Up!: Impact of a Quality Improvement Intervention to Promote Early Mobilization in Critically Ill Children. Pediatr Crit Care Med. 2016 Dec;17(12):e559-e566. doi: 10.1097/PCC.0000000000000983. PMID 27759596
- [Background] Miura S, Wieczorek B, Lenker H, Kudchadkar SR. Normal Baseline Function Is Associated With Delayed Rehabilitation in Critically Ill Children. J Intensive Care Med. 2020 Apr;35(4):405-410. doi: 10.1177/0885066618754507. Epub 2018 Jan 22. PMID 29357778
- [Background] Pun BT, Balas MC, Barnes-Daly MA, Thompson JL, Aldrich JM, Barr J, Byrum D, Carson SS, Devlin JW, Engel HJ, Esbrook CL, Hargett KD, Harmon L, Hielsberg C, Jackson JC, Kelly TL, Kumar V, Millner L, Morse A, Perme CS, Posa PJ, Puntillo KA, Schweickert WD, Stollings JL, Tan A, D'Agostino McGowan L, Ely EW. Caring for Critically Ill Patients with the ABCDEF Bundle: Results of the ICU Liberation Collaborative in Over 15,000 Adults. Crit Care Med. 2019 Jan;47(1):3-14. doi: 10.1097/CCM.0000000000003482. PMID 30339549
- [Derived] Azamfirei R, Behrens D, Padilla S, Madden K, Goldberg S, Geno M, Manning MJ, Piole M, Madsen E, Maue D, Abu-Sultaneh S, Awojoodu R, Wang NY, Needham DM, Neufeld K, Kudchadkar SR. Delirium Screening in Critically Ill Children: Secondary Analysis of the Multicenter PICU Up! Pilot Trial Dataset, 2019-2020. Pediatr Crit Care Med. 2024 Oct 1;25(10):880-888. doi: 10.1097/PCC.0000000000003555. Epub 2024 Jun 4. PMID 38832837